CLINICAL TRIAL: NCT05399368
Title: A Phase 2 Study to Evaluate the Efficacy and Safety of RPT193 as Monotherapy in Adults With Moderate-to-Severe Atopic Dermatitis
Brief Title: An Efficacy and Safety Study of RPT193 in Adults With Atopic Dermatitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study on clinical hold by FDA
Sponsor: RAPT Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RPT193-02
Record Dates: First submitted 2022-05-26; First posted 2022-06-01 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Atopic Dermatitis
Keywords: atopic dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- RPT193 400 mg (Experimental): RPT193 400 mg oral tablet administered daily for 16 weeks
  Interventions: Drug: RPT193
- RPT193 200 mg (Experimental): RPT193 200 mg oral tablet administered daily for 16 weeks
  Interventions: Drug: RPT193
- RPT193 50 mg (Experimental): RPT193 50 mg oral tablet administered daily for 16 weeks
  Interventions: Drug: RPT193
- Placebo (Placebo Comparator): Matching placebo oral tablet administered daily for 16 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: RPT193 — RPT193 is an antagonist of the C-C motif chemokine receptor 4 (CCR4) that inhibits CCR4-mediated chemotaxis toward both CCL22 and CCL17
  Arms: RPT193 200 mg; RPT193 400 mg; RPT193 50 mg
Other: Placebo — Nonactive placebo tablet
  Arms: Placebo

SUMMARY:
Phase 2 study of RPT193 in adults with atopic dermatitis

DETAILED DESCRIPTION:
Randomized, placebo-controlled Phase 2 study of RPT193 in adults with moderate-to-severe atopic dermatitis

ELIGIBILITY:
Inclusion Criteria:

* Clinically confirmed diagnosis of active atopic dermatitis (AD), according to the revised Hanifin and Rajka criteria
* 12-month history of AD and had no significant flares in AD for at least 4 weeks before screening
* inadequate response to a ≥1 month treatment with topical medications
* Atopic dermatitis covering ≥10% of the body surface area
* EASI score ≥16
* Validated Investigator Global Assessment (VIGA) ≥3
* Use of emollient(s) at least 2x daily for 1 week prior to baseline
* Negative coronavirus disease (COVID)-19 results at screening

Exclusion Criteria:

* Uncontrolled moderate-to-severe asthma
* Uncontrolled diabetes
* Stage III or IV cardiac failure
* Severe renal condition
* Major surgery within 8 weeks of screening
* Immunodeficiency and/or receipt of immunosuppressive drugs within 4 weeks of baseline
* Use of systemic Janus kinase (JAK) inhibitor within 8 weeks of baseline
* Received live or live-attenuated vaccine within 4 weeks of baseline
* Prior receipt of RPT193

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-05-24 (Actual)

PRIMARY OUTCOMES:
Clinical efficacy | 16 weeks
  % change in Eczema Area Severity Index (EASI)
Safety as measured by adverse events | 16 weeks
  Incidence of treatment-emergent adverse events

CONTACTS AND LOCATIONS:
Locations (59):
- United States (56):
  - Cahaba Dermatology and Skin Health Center, Birmingham, Alabama
  - Perseverance Research Center, Scottsdale, Arizona
  - Arkansas Research Trials, LLC, North Little Rock, Arkansas
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - First OC Dermatology, Fountain Valley, California
  - Grimes Center, Los Angeles, California
  - Dermatology Research Associates, Los Angeles, California
  - Wallace Medical Group, Los Angeles, California
  - Velocity Clinical Research, North Hollywood, California
  - Integrative Skin Science and Research, Sacramento, California
  - Clinical Science Institute, Santa Monica, California
  - Clinical Trials Research Institute, Thousand Oaks, California
  - Foxhall Research Center, Washington D.C., District of Columbia
  - Driven Research LLC, Coral Gables, Florida
  - Florida Academic Centers Research and Education, LLC, Coral Gables, Florida
  - Palm Beach Dermatology Group, Delray Beach, Florida
  - GSI Clinical Research, Margate, Florida
  - Lenus Research & Medical Group, LLC, Sweetwater, Florida
  - Forcare Clinical Research, Tampa, Florida
  - Skin Care Physicians of Georgia, Macon, Georgia
  - Marietta Dermatology Clinical Research, Inc., Marietta, Georgia
  - Georgia Skin & Cancer Clinic, Savannah, Georgia
  - University Dermatology and Vein Clinic, Darien, Illinois
  - Indiana Clinical and Translational Sciences Institute (CTSI) Clinical Research Center, Indianapolis, Indiana
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - The Indiana Clinical Trials Center PC, Plainfield, Indiana
  - Skin Sciences PLLC, Louisville, Kentucky
  - DelRicht Research, Baton Rouge, Louisiana
  - Schweiger Dermatology Group, PC Research Division, Columbia, Maryland
  - MetroBoston Clinical Partners, Brighton, Massachusetts
  - Beacon Clinical Research, LLC, Quincy, Massachusetts
  - Fivenson Dermatology, Ann Arbor, Michigan
  - St. Joseph Dermatology and Vein Clinic, Saint Joseph, Michigan
  - Grekin Skin Institute, Warren, Michigan
  - Medisearch Clinical Trials, Saint Joseph, Missouri
  - Advanced Dermatology of the Midlands, Omaha, Nebraska
  - Skin Specialists PC (Schlessinger MD), Omaha, Nebraska
  - Schweiger Dermatology Group, Verona, New Jersey
  - Forest Hills Dermatology Group, Kew Gardens, New York
  - JUVA Skin & Laser Center, New York, New York
  - Ichan School of Medicine at Mount Sinai, New York, New York
  - Markowitz Medical, PLLC, New York, New York
  - Optima Research - Boardman, Boardman, Ohio
  - Apex Clinical Research Center, Mayfield Heights, Ohio
  - Health Concepts, Rapid City, South Dakota
  - Arlington Research Center Inc., Arlington, Texas
  - DermResearch, Austin, Texas
  - Studies in Dermatology, LLC, Cypress, Texas
  - Dermatology Treatment and Research Center, Dallas, Texas
  - Clinical Trial Network, Houston, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - Acclaim Dermatology, Sugar Land, Texas
  - Complete Dermatology, Sugar Land, Texas
  - Jordan Valley Dermatology Center, South Jordan, Utah
  - West End Dermatology Associates, Richmond, Virginia
  - Premier Clinical Research, Spokane, Washington
- Canada (3):
  - SimcoDerm Medical and Surgical Dermatology Center, Barrie, Ontario
  - LEADER Research, Hamilton, Ontario
  - Red Maple Trials Inc., Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No